CLINICAL TRIAL: NCT04973319
Title: Trastuzumab Combined With Pertuzumab and Sequential Use of Pyrotinib vs. Trastuzumab Combined With Pertuzumab for Adjuvant Treatment of Breast Cancer After Neoadjuvant Therapy
Brief Title: Trastuzumab Combined With Pertuzumab for Adjuvant Treatment of Breast Cancer After Neoadjuvant Therapy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Director, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shengjing-LCG008
Record Dates: First submitted 2021-07-07; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; pyrotinib; trastuzumab; pertuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Trastuzumab; pertuzumab

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Each subject in the test group will receive the test drug (pyrotinib) for 52 weeks, and will be followed up for at least 3 years from the start of randomization, until disease recurrence, intolerable toxicity, withdrawal of informed consent, or termination of the medication as per the investigator's judgment. The subject who has a second primary malignant tumor in a non-breast area will continue to be followed up until a recurrent disease or death due to primary breast cancer. The subjects who are hormone receptor-positive will be advised to receive endocrinotherapy simultaneously. Within 28 days after the last administration of the test drug, the subjects in the test group must complete the safety follow-up and the end-of-treatment visit and continue to receive the follow-up visit.
  Interventions: Drug: Pyrotinib
- control group (Other): Each enrolled subject will complete at least ≥ 24 weeks (8 drug delivery cycles) of trastuzumab combined with pertuzumab in the neoadjuvant and/or adjuvant treatment phase.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Pyrotinib — Each subject in the test group will receive the test drug (pyrotinib) for 52 weeks, and will be followed up for at least 3 years from the start of randomization, until disease recurrence, intolerable toxicity, withdrawal of informed consent, or termination of the medication as per the investigator's judgment.
  Other Names: Trastuzumab and pertuzumab
  Arms: test group
Drug: Trastuzumab — Each enrolled subject will complete at least ≥ 24 weeks (8 drug delivery cycles) of trastuzumab combined with pertuzumab in the neoadjuvant and/or adjuvant treatment phase.
  Other Names: pertuzumab
  Arms: control group

SUMMARY:
Patients with HER-2 positive breast cancer who have poor outcomes after endocrinotherapy and standard chemotherapy can be significantly improved by the use of anti-HER-2 monoclonal antibody trastuzumab. In the current clinical practice of neoadjuvant therapy, trastuzumab combined with chemotherapy can significantly increase the pCR and improve the outcomes in patients. However, there seems to be no available treatment for patients who have no pCR and still have residual tumors except for sequential trastuzumab treatment for 1 year. Compared with trastuzumab, a HER-2 macromolecule inhibitor, pyrotinib has a different site of action and an increased EGFR target. Compared with lapatinib, a small molecule inhibitor of EGFR and HER-2, pyrotinib is an irreversible inhibitor, with the ability to achieve a better curative effect at a lower human plasma exposure level. This trial is designed to evaluate the effectiveness and safety of trastuzumab combined with pertuzumab followed by sequential pyrotinib treatment in non-pCR patients after neoadjuvant therapy.

DETAILED DESCRIPTION:
In recent years, the interest has greatly increased in how to proceed with postoperative intensive adjuvant therapy for early breast cancer patients who have not reached pCR and still have residual lesion after neoadjuvant therapy. Relevant efficacy and safety data have been continuously verified in clinical trials, and some treatments have been clinically approved. Moreover, new attempts and explorations are still going on in clinical practice. Based on the preliminary clinical findings, it is planned to design a randomized controlled, open-label, multi-center phase III clinical study that will explore the efficacy of trastuzumab combined with pertuzumab for 1 year followed by sequential pyrotinib vs. touzumab combined with pertuzumab for 1 year, aiming to verify that dual-target adjuvant therapy with sequential use of pyrotinib maleate tablets is superior to dual-target adjuvant therapy alone in HER-2 positive early breast cancer patients who have not reached pCR after neoadjuvant therapy. If this clinical trial achieves a positive result, the use of pyrotinib maleate tablets will be promoted for early breast cancer patients who have not reached pCR and still have residual tumor lesions after neoadjuvant therapy with an attempt to further achieve improved outcomes and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 but ≤ 75 years (The maximal age of the subjects enrolled in the Phase 3 study of pyrotinib is 75 years old, and there is no safety data for the use of the drug in older people);
* ECOG level 0-1;
* Primary infiltrating breast lesions and lymph nodes should follow these conditions at the same time: histologically confirmed invasive breast cancer; receiving neoadjuvant treatment and completing the operation, with postoperative pathological examination indicating residual invasive cancer in the breast or axillary lymph nodes; HER2-positive breast cancer is confirmed in the pathology test, with 3+ in immunohistochemistry (IHC) test and HER2 gene amplification (HER2/CEP17 ≥ 2.0 or average HER2 copy number/cell number ≥ 6); no recurrent and metastatic disease after surgery;
* HER-2 positive breast cancer patients who have non-pCR after trastuzumab+pertuzumab as neoadjuvant therapy, and have completed trastuzumab combined with pertuzumab as adjuvant treatment. During the neoadjuvant and/or adjuvant therapy phase, at least ≥24 weeks (8 drug delivery cycles) of trastuzumab + pertuzumab. And the time interval from the end of the last trastuzumab treatment to entering the trial must be ≤ 1 year;
* Hormone receptor status (ER and PR) that is known;
* The functional level of major organs must conform to the following requirements (no blood transfusion, no use of white blood cell- and platelet-increasing drugs within 2 weeks before screening): Neutrophils (ANC) ≥ 1.5×109/L; Platelet count (PLT) ≥ 90×109/L; Hemoglobin (Hb) ≥ 90 g/L; Total bilirubin (TBIL)≤ 1.5×upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5×ULN;
* Female patients who are not menopausal or not surgically sterilized agree to abstain from sex or use effective non-hormonal drugs for contraception during the treatment period and within 8 weeks after the last administration;
* Patients who participate in the trial voluntarily, sign an informed consent, have good compliance and are willing to comply with the follow-up visit.

Exclusion Criteria:

* With a history of recurrent local or regional breast disease;
* Stage IV (metastatic) breast cancer;
* Bilateral breast cancer;
* With a history of any malignancies other than breast cancer in the past 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or squamous cell carcinoma;
* Patients who have received pyrotinib, lapatinib, neratinib or other tyrosine kinase inhibitors, enmetrastuzumab (T-DM1), and other anti-tumor biological therapies or tumor immunotherapy;
* Patients who are receiving anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy or immunotherapy;
* Severe heart disease or discomfort, including but not limited to the following diseases: a confirmed history of heart failure or systolic dysfunction (LVEF < 50%); high-risk uncontrolled arrhythmia, such as atrial tachycardia, remarkable ventricular arrhythmia (such as ventricular tachycardia) or higher-grade atrioventricular block; angina pectoris requiring anti-angina medication; clinically significant valvular disease; transmural myocardial infarction shown by ECG; uncontrolled blood pressure in patients with hypertension who have been given antihypertensive drugs (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg);
* Inability to swallow, intestinal obstruction or other factors that affect drug taking and absorption;
* With a history of diagnosed neurological or mental disorders, including involuntary behavior or mental illness;
* With a history of gastrointestinal diseases with diarrhea as the main symptom;
* Patients who are known to have a history of allergies to the drug components in this trial; have a history of immunodeficiency, including HIV positive results, or other acquired or congenital immunodeficiency diseases; or have a history of organ transplantation;
* Female patients during pregnancy and lactation, or those who are fertile and positive for baseline pregnancy test;
* Serious concomitant diseases or other comorbid diseases that will interfere with the planned treatment, including infectious diseases with active infections (including but not limited to hepatitis B, active hepatitis C, active tuberculosis, active syphilis, etc.); or any other cases in which the investigator believes that the patient cannot participate in the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 450 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (IDFS) | at least 3 years from the beginning of randomization.
  the time from the date of randomization to the first appearance of recurrent disease. Recurrent diseases include ipsilateral or contralateral breast cancer, local or regional recurrence, distant recurrence and death from any cause.

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | at least 3 years from the date of randomization
  the time from the date of randomization to the first occurrence of any recurrent disease. Recurrent diseases include second primary malignant tumor in the non-breast region and preinvasive cancer in the breast duct.
overall survival (OS) | at least 3 years from the date of randomization
  the time from the date of randomization to death due to any cause.
Distant Disease-Free Survival (DDFS) | at least 3 years from the date of randomization
  the time from the date of randomization to the first occurrence of distant recurrence or death from any cause

OTHER OUTCOMES:
Adverse event (AE) | from the date of randomization to no more than 28 days after the last drug withdrawal.
  AEs will be assessed as per the NCI-CTC AE 5.0 standard.

CONTACTS AND LOCATIONS:
Overall Officials: Cai-Gang Liu, MD, Principal Investigator — Department of Breast Surgery, Shengjing Hospital affiliated to China Medical University
Locations (1):
- Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No